CLINICAL TRIAL: NCT05158283
Title: Clinical Of Chocolate Balloon Dilatation Versus Plain Balloon Dilatation to Treat Arteriosclerosis Occlusive Disease of Lower Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH202109
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Atherosclerosis; Ischemia
Keywords: Chocolate balloon; infrapopliteal artery
MeSH Terms: conditions — Atherosclerosis; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Chocolate balloon (Experimental): Chocolate balloon group
  Interventions: Device: chocolate balloon
- Intervention: plain balloon (Experimental): plain balloon group
  Interventions: Device: plain balloon

INTERVENTIONS:
Device: chocolate balloon — chocolate balloon dilatation
  Arms: Intervention: Chocolate balloon
Device: plain balloon — plain balloon dilatation
  Arms: Intervention: plain balloon

SUMMARY:
This is a Prospective randomized controlled study to evaluate the difference of safety，effectiveness between chocolate balloon and plain balloon dilatation in treatment of infrapopliteal artery lesions.

DETAILED DESCRIPTION:
Prospective randomized controlled study to evaluate the difference of safety，effectiveness between chocolate balloon and plain balloon dilatation in treatment of infrapopliteal artery lesions. Patients with femoral-popliteal artery lesions in our department were randomly assigned to the chocolate balloon group and plain balloon dilatation group. Compare the ischemic improvement rate (limb salvage rate, postoperative patency rate) and the complications rate of two different treatments.

ELIGIBILITY:
Inclusion criteria： 1.all patients signed an informed consent form; 2.digital subtraction angiography (DSA) revealed femoropopliteal artery stenosis above 70% or occlusion resulting in claudication (Rutherford clinical category-Becker class II-III2-3) or critical limb ischemia (CLI) (Rutherford clinical category 4-5-Becker class IV-V) 3.with unobstructed vascular inflow; 4.with at least a vessel runoff; 5. good compliance and regular follow-up.

Exclusion criteria: 1. Acute or subacute lower limb ischemia caused by acute intraluminal thrombus within the target lesion.; 2. Severe calcified lesions （grade 4 in the PACSS scale）; 3. In-stent restenosis lesion or surgical arterial bypass grafting; 4. Severe renal insufficiency: creatinine level greater than 2.5 mg/dL; 5. Platelet count below 100,000/μL or with antiplatelet / anticoagulation contraindications; 6. Immunologic diseases or malignant diseases; 7. Ongoing active infection; 8. Decompensated congestive heart failure or acute coronary syndrome; 9. Refuse to sign the informed consent Unwillingness to comply with follow-up suggestions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success rate | 1 day
  Technical success was defined as residual stenosis less than 30% by final
freedom from clinically-driven TLR rate | 12 months
  it is defined as thefreedom from clinically-driven target lesion revascularization
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization , and significant embolic events, which were defined as causing end-organ damage.
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided